CLINICAL TRIAL: NCT05416983
Title: The Development of a Shared Decision-Making Encounter Tool for Decisions of Adjuvant Treatment in Patients With Resected Non-Small Cell Lung Cancer
Brief Title: Developing a Shared Decision Making Tool for Patients With Surgically Removed Non-small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 21-013359; NCI-2022-01685 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-06-06; First posted 2022-06-14 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Lung Non-Small Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (discussion): Patient and clinician discussions are observed to support refinement of a decision aid. Clinicians may use a prototype of the decision aid in discussions with their patients and may complete a questionnaire.
  Interventions: Procedure: Discussion; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Discussion — Attend discussion
Other: Questionnaire Administration — Complete questionnaire

SUMMARY:
This study observes conversations between non-small cell lung cancer patients and their doctors to support the development of a decision aid that can be used to inform discussions about treatment options for after surgery. Patients who have undergone surgery for their non-small cell lung cancer may have the option of completing additional treatment. Patients contemplating this additional treatment have been shown to be most satisfied with their choice if they perceive an effort by their doctor to share decision making. Shared decision making tools can help doctors guide conversations, offer tailored recommendations, and support deliberation on whether or not to pursue treatment. This study develops a shared decision making tool for patients with surgically removed non-small cell lung cancer contemplating additional treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To develop, in close collaboration with stakeholders, an evidence-based decision aid to inform discussions regarding options for adjuvant treatment in patients with resected non-small cell lung cancer (NSCL) (NSCL adjuvant choice).

OUTLINE:

Patient and clinician discussions are observed to support refinement of a decision aid. Clinicians may use a prototype of the decision aid in discussions with their patients and may complete a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS:
* Adults >= 18 years with biopsy proven resected non-small cell lung cancer (NSCLC)
* Appointments to discuss adjuvant treatment of resected NSCLC
* CLINICIANS:
* Clinicians who meet with patients to discuss adjuvant treatment of resected NSCLC
* PAG MEMBERS:
* Adults >= 18 years
* Member of the Knowledge and Evaluation Research (KER) Unit Patient Advisory Group (PAG)

Exclusion Criteria:

* PATIENTS
* Major barriers to providing informed consent (i.e., dementia, severe hearing or visual impairment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with resected non-small cell lung cancer, clinicians, and PAG members.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Development of decision aid | Up to study completion, up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Leventakos, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials